CLINICAL TRIAL: NCT06068270
Title: Randomized Clinical Trial on the Effect of Micro-osteoperforations (MOPs) During Intrusion of Flared Upper Anterior Teeth in Stage IV Periodontitis Patients
Brief Title: Effect of MOPs During Orthodontic Movement in Periodontitis Patients
Acronym: MOPorthoperi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Concepción Martín Alvaro, Professor in Orthodontics, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URI_113-210923
Record Dates: First submitted 2023-09-21; First posted 2023-10-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Stage IV Periodontitis; Orthodontic Tooth Movement
Keywords: Stage IV periodontitis; Orthodontic tooth movement; Micro-osteoperforations
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Comparative 2-arm parallel single-blinded randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): According to randomization, test group patients will receive MOPs at the beginning of the orthodontic therapy and at every other orthodontic recall appointment.
  Interventions: Procedure: Micro-ostoperforations (MOPs)
- Control group (No Intervention): No MOPs performed at any stage of the orthodontic therapy

INTERVENTIONS:
Procedure: Micro-ostoperforations (MOPs) — 3 MOPs will be performed in the bone next to the root of the experimental tooth. MOPs will be performed using the Excellerator® (Propel Orthodontics, Denstply, Sirona)
  Arms: Test group

SUMMARY:
Micro-osteoperforations (MOPs) cause cortical bone injuries and consequently increase the expression of inflammatory mediators, allowing for increased bone and periodontal ligament remodeling associated with orthodontic movement. It remains unclear the effect of orthodontic intrusion combined with MOPs application on teeth with reduced periodontium. The general objective will be to determine the efficacy of MOPs during orthodontic tooth movement (OTM) in terms of periodontal and orthodontic outcomes in stage IV periodontitis patients, case type 2 with pathological tooth migration (PTM), characterized the presence of at least one flared tooth of the upper-anterior sextant with an intrabony defect (intrabony component <5mm)

DETAILED DESCRIPTION:
This is a comparative 2-arm parallel single-blinded randomized controlled clinical trial, with allocation ratio of 1:1, aimed to test an intervention (the use of MOPs) on CAL changes 12 months after placing orthodontic appliances. The control intervention will be the same treatment without the bone traumatic intervention.

Sample: Patients with stage IV periodontitis case type 2 characterized with PTM characterized the presence of at least one flared tooth of the upper-anterior sextant with an intrabony defect (intrabony component <5mm) attending the Post-graduate Program of Periodontology and the Post-graduate Program of Orthodontics of the Faculty of Dentistry at the Complutense University of Madrid (UCM).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if agreeing to undertake combined periodontal and orthodontic therapy following the clinical practice guideline of stage IV periodontitis patients, and fulfilling the following criteria:

* adult patients older than 18-year-old;
* systemically healthy (see exclusion criteria);
* diagnosed as stage IV (Papapanou et al., 2018) case-type 2 (Herrera et al. 2022) periodontitis;
* the presence of at least one flared tooth of the upper-anterior sextant with an intrabony defect (intrabonny component <5mm) (experimental teeth);
* in need of orthodontic therapy.

Exclusion Criteria:

* systemic diseases (diabetes mellitus, obesity, cardiovascular diseases);
* any medication that could affect the level of inflammation, (such as chronic antibiotics, phenytoin, cyclosporin, anti-inflammatory drugs, systemic corticosteroids, or calcium channel blockers);
* pregnant or lactating woman;
* inability to respond questions or to attend follow-up visits;
* extreme skeletal malocclusions requiring orthognathic surgery;
* patients smoking more than 10 cigarettes/day; and
* the presence of PD greater or equal to 5mm with BOP after step 3 of periodontal therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
CAL | 12 months
  clinical attachment level (CAL) in mm

SECONDARY OUTCOMES:
Type of movement | 12 months
  Description of the type of movement (categorical outcome)
Duration of orthodontic treatment | >12 months
  Total duration in months
External apical root resorption (EARR) | 12 months
  Presence of EARR (in mm3)
Probing pocket depth (PPD) | 12 months
  PPD in mm
Gingival margin level (GM) | 12 months
  GM in mm
Gingival recessions | 12 months
  Recessions in mm
Bleeding on probing (BOP) | 12 months
  BOP (presence or absence)
Suppuration on probing (SOP) | 12 months
  SOP (presence or absence)
Plaque index (PI) | 12 months
  PI (categorical outcome)
Radiographic periodontal outcomes | 12 months
  Radiographic bone level (RBL), radiographic defect angle
Inflammatory biomarkers in gingival crevicular fluid (GCF) | 12 months
  Inflammatory biomarkers RANKL and OPG, in picograms.
Oral health related quality of life questionnaire (OHRQoL) | 12 months
  Oral health related quality of life questionnaire (OHRQoL)
Pain questionnaire | 12 months
  Pain questionnaire (VAS scale 0-100)
Aesthetic component of the Index of Orthodontic Treatment Need (IOTN) | 12 months
  IOTN after orthodontic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Conchita Martin, Prof, Principal Investigator — Universidad Complutense de Madrid; Elena Figuero, Prof, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Faculty of Odontology, University Complutense Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available